CLINICAL TRIAL: NCT01370525
Title: A Phase III Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial of 14 Day Treatment With Esomeprazole 20 mg Once Daily in Subjects With Frequent Heartburn
Brief Title: Efficacy of Esomeprazole in Patients With Frequent Heartburn
Acronym: NEXT1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D961RC00001
Record Dates: First submitted 2011-06-01; First posted 2011-06-10 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-02

CONDITIONS: Heartburn
Keywords: Heartburn
MeSH Terms: conditions — Heartburn | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Esomeprazole 20 mg (Experimental)
  Interventions: Drug: Esomeprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Nexium 20 mg administered as 22.3 mg of esomeprasole magnesium hydrate, capsule, oral dose

SUMMARY:
This study will investigate the efficacy of esomeprazole 20 mg once a day in the treatment of frequent heartburn

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant ,non-lactating females 18 years or older
* Experience heartburn at least 2 days a week
* Having heartburn that has responded to heartburn medication
* Must discontinue any current heartburn medications

Exclusion Criteria:

* Having a history of erosive esophagitis verified by endoscopy
* Having a history of GERD which was diagnosed by a physician
* Inability to take study medication or complete the study and all study procedures
* Subjects that have required more than one 14-day course of PPI treatment within the past 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tore Lind, MD, Study Director — AstraZeneca
Locations (10):
- United States (10):
  - Research site, Sacramento, California
  - Research site, Seminole, Florida
  - Research site, Meridian, Idaho
  - Research site, Indianapolis, Indiana
  - Research site, Metairie, Louisiana
  - Research site, Omaha, Nebraska
  - Research site, Raleigh, North Carolina
  - Research site, Cleveland, Ohio
  - Research site, Mt. Pleasant, South Carolina
  - Research site, San Antonio, Texas

REFERENCES:
- [Derived] Peura D, Le Moigne A, Wassel H, Pollack C. Analysis of the symptom response to esomeprazole 20 mg over days 1-4 of a 14-day course of treatment for frequent heartburn: results of two randomised controlled trials. BMJ Open Gastroenterol. 2019 Jun 21;6(1):e000278. doi: 10.1136/bmjgast-2019-000278. eCollection 2019. PMID 31297231
- [Derived] Peura DA, Le Moigne A, Wassel H, Pollack C. Sustained efficacy following resolution of frequent heartburn with an over-the-counter regimen of esomeprazole 20 mg or placebo for 14 days: two randomized trials. BMC Gastroenterol. 2018 May 22;18(1):69. doi: 10.1186/s12876-018-0790-2. PMID 29788903
- [Derived] Peura D, Le Moigne A, Pollack C, Nagy P, Lind T. A 14-day regimen of esomeprazole 20 mg/day for frequent heartburn: durability of effects, symptomatic rebound, and treatment satisfaction. Postgrad Med. 2016 Aug;128(6):577-83. doi: 10.1080/00325481.2016.1203236. Epub 2016 Jul 4. PMID 27331882
- [Derived] Peura DA, Traxler B, Kocun C, Lind T. Esomeprazole treatment of frequent heartburn: two randomized, double-blind, placebo-controlled trials. Postgrad Med. 2014 Jul;126(4):33-41. doi: 10.3810/pgm.2014.07.2781. PMID 25141241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From total of 486 enrolled subjects, 340 subjects were randomised. From 340 subjects 171 and 169 were allocated to Esomeprazole and Placebo respectively.
Groups:
- Esomeprazole: Nexium 20 mg administered as 22.3 mg of esomeprasole magnesium hydrate
- Placebo: Placebo for Esomeprazole
Period: Overall Study
Arm/Group | Esomeprazole | Placebo
Started | 171 | 169
Patients Who Received Treatment | 168 | 163
Patients Who Completed Treatment | 163 | 158
Completed | 163 | 158
Not Completed | 8 | 11
Not completed — Voluntary Discontinuation by Subject | 2 | 3
Not completed — Eligibility criteria not fulfilled | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to follow up | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Esomeprazole: Esomeprazole magnesium trihydrate 22.3 mg
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Placebo | Total
Number analyzed (Participants) | 171 | 169 | 340
Age Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (12.2) | 45.9 (12.6) | 44.75 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 97 | 202
  Male | 66 | 72 | 138
Race/Ethnicity, Customized [Number; unit: Participants] — Randomized population was analyzed using criteria of white/ black or african american/ asian/ american indian or alaska native /white.
  Participants
    WHITE | 103 | 112 | 215
    BLACK OR AFRICAN AMERICAN | 65 | 55 | 120
    ASIAN | 0 | 1 | 1
    AMERICAN INDIAN/ALASKA NATIVE | 1 | 0 | 1
    OTHER | 2 | 1 | 3
Race/Ethnicity, Customized [Number; unit: Participants] — Randomized population was analyzed using criteria of hispanic or latino/ not hispanic or latino/ not reported.
  Participants
    HISPANIC OR LATINO | 34 | 26 | 60
    NOT HISPANIC OR LATINO | 56 | 59 | 115
    NOT REPORTED | 81 | 84 | 165

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heartburn Free 24 Hour Days During 14 Days of Randomized Treatment
Time Frame: From randomisation to day 14
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 168 | 163
Percentage | 43.32 (34.36) | 29.44 (29.83)

2. Secondary Outcome: Number of Subjects Reporting Heartburn 2 Days or Less During the 14 Days Randomized Treatment Period
Description: Randomized treatment period is considered as both weeks 1 and 2 between V3 and V4.
Time Frame: From randomisation to day 14
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 168 | 163
Participants | 27 | 7

3. Secondary Outcome: Comparison of Number of Subjects With 0, 1, 2, 3 or 4 Days With no Heartburn Over Days 1 to 4 Between Esomeprazole 20 mg and Placebo
Description: The first 4 consecutive days subjects were on randomized treatment, between V3 and V4.
Time Frame: From randomisation to the day 14
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 168 | 163
Participants
  Zero days | 64 | 76
  One day | 25 | 36
  Two days | 36 | 18
  Three days | 25 | 21
  Four days | 18 | 12

4. Secondary Outcome: Number of Subjects With Heartburn 1 Day or Less During the Final Week, Second Week, First Week of Treatment
Description: There were three separate 7 day time periods during the treatment period; The first week (days 1-7), the second week (days 8-14), and the last 7 consecutive days (last day subject reported and the prior 6). For a given subject, the second week and last 7 consecutive days are the same if the subject has recorded measurements for the entire 14 day treatment period. However, for subjects reporting anything less than 14 days the two will not be identical. For all three 7 day time periods, days when a subject did not call in (i.e., missing values) were imputed as a day with heartburn.
Time Frame: From randomisation to day 14
Measure: Number; unit: Participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 168 | 163
Participants
  Last 7 consecutive days | 43 | 17
  Second 7 calender days | 43 | 16
  First 7 calendar days | 26 | 10

5. Primary Outcome: Percentage of Heartburn Free 24 Hour Days During 14 Days of Randomized Treatment
Time Frame: From randomization to day 14
Population: Per-protocol analysis set
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 150 | 149
Percentage | 44.52 (34.4) | 31.25 (30.26)

ADVERSE EVENTS:
Description: Full analysis set (FAS) population was analyzed.
Arm/Group | Esomeprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/163
Other Adverse Events (participants affected / at risk) | 18/168 | 15/163
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole (N=168) | Placebo (N=163)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 5 | 3
Diarhhoea (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Headache (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days